CLINICAL TRIAL: NCT01989676
Title: A PHASE 3 RANDOMIZED, DOUBLE-BLIND STUDY OF PF-05280014 PLUS PACLITAXEL VERSUS TRASTUZUMAB PLUS PACLITAXEL FOR THE FIRST-LINE TREATMENT OF PATIENTS WITH HER2-POSITIVE METASTATIC BREAST CANCER
Brief Title: A Study Of PF-05280014 [Trastuzumab-Pfizer] Or Herceptin® [Trastuzumab-EU] Plus Paclitaxel In HER2 Positive First Line Metastatic Breast Cancer Treatment (REFLECTIONS B327-02)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B3271002; REFLECTIONS B327-02; 2013-001352-34 (EudraCT Number); B3271002 (Other: Alias Study Number)
Record Dates: First submitted 2013-10-28; First posted 2013-11-21 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Metastatic Breast Cancer
Keywords: Phase 3; trastuzumab; Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — PF-05280014; Paclitaxel; Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PF-05280014 (Experimental)
  Interventions: Biological: PF-05280014; Drug: Paclitaxel
- Herceptin® (Active Comparator)
  Interventions: Biological: Herceptin®; Drug: Paclitaxel

INTERVENTIONS:
Biological: PF-05280014 — Concentrate for solution for infusion, sterile vial 150 mg. Initial dose of 4 mg/kg over 90 minutes (depending on tolerability) IV infusion, then 2 mg/kg over 30 to 90 minutes (depending on tolerability) IV infusion until disease progression. Following completion of the paclitaxel administration period and beginning no earlier than Week 33 of the study, the PF-05280014 regimen may be changed at the discretion of the investigator to every 3 weeks at a dose of 6 mg/kg infused over 30 to 90 minutes depending on tolerability.
  Other Names: Trastuzumab-Pfizer
  Arms: PF-05280014
Drug: Paclitaxel — A nonaqueous solution intended for dilution with a suitable parenteral fluid prior to intravenous infusion. Paclitaxel is available in 30 mg (5 mL), 100 mg (16.7 mL), and 300 mg (50 mL) multidose vials. Each mL of sterile nonpyrogenic solution contains 6 mg paclitaxel. The starting dose of paclitaxel will be 80 mg/m^2 by IV infusion over 60 minutes (duration of infusion may be modified according to local standard of care, if applicable). Provision is made for dose reduction to 70 mg/m^2 and then 60 mg/m^2 as needed. In the absence of disease progression in the judgment of the investigator or prohibitive toxicity, patients will receive treatment with paclitaxel for at least 6 cycles or until maximal benefit of response is obtained, in the judgment of the investigator.
  Arms: PF-05280014
Biological: Herceptin® — Concentrate for solution for infusion, sterile vial 150 mg. Initial dose of 4 mg/kg over 90 minutes (depending on tolerability) IV infusion, then 2 mg/kg over 30 to 90 minutes (depending on tolerability) IV infusion weekly until disease progression. Following completion of the paclitaxel administration period and beginning no earlier than Week 33 of the study, the Herceptin® regimen may be changed at the discretion of the investigator to every 3 weeks at a dose of 6 mg/kg infused over 30 to 90 minutes depending on tolerability.
  Other Names: Trastuzumab (EU)
  Arms: Herceptin®
Drug: Paclitaxel — A nonaqueous solution intended for dilution with a suitable parenteral fluid prior to intravenous infusion. Paclitaxel is available in 30 mg (5 mL), 100 mg (16.7 mL), and 300 mg (50 mL) multidose vials. Each mL of sterile nonpyrogenic solution contains 6 mg paclitaxel. The starting dose of paclitaxel will be 80 mg/m^2 by IV infusion over 60 minutes (duration of infusion may be modified according to local standard of care, if applicable). Provision is made for dose reduction to 70 mg/m^2 and then 60 mg/m^2 as needed. In the absence of disease progression in the judgment of the investigator or prohibitive toxicity, patients will receive treatment with paclitaxel for at least 6 cycles or until maximal benefit of response is obtained, in the judgment of the investigator.
  Arms: Herceptin®

SUMMARY:
The current study will compare the efficacy, safety, pharmacokinetics and immunogenicity of PF-05280014 in combination with paclitaxel versus trastuzumab sourced from the European Union (trastuzumab-EU) with paclitaxel in female patients with HER2-positive, metastatic breast cancer in the first-line treatment setting. The hypothesis to be tested in this study is that the efficacy (ORR) of PF-05280014 is similar to trastuzumab-EU.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of breast cancer.
* Presence of metastatic disease.
* Documentation of HER2 gene amplification or overexpression.
* Available tumor tissue for central review of HER2 status.
* At least 1 measurable lesion as defined by RECIST 1.1.
* Eastern Cooperative Oncology Group status of 0 to 2.
* Left ventricular ejection fraction within institutional range of normal, measured by either two dimensional echocardiogram or multigated acquisition scan.

Exclusion Criteria:

* Relapse within 1 year of last dose of previous adjuvant (including neoadjuvant) treatment (except endocrine therapy) and within 1 year before randomization.
* Prior systemic therapy for metastatic disease (except endocrine therapy).
* Prior cumulative dose of doxorubicin of >400 mg/m2, epirubicin dose >800 mg/m^2, or the equivalent dose for other anthracyclines or derivatives (eg, 72 mg/m^2 of mitoxantrone). If the patient has received more than one anthracycline, then the cumulative dose must not exceed the equivalent of 400 mg/m^2 of doxorubicin.
* Inflammatory breast cancer.
* Active uncontrolled or symptomatic central nervous system metastases.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 707 (Actual)
Dates: Start 2014-02-24 (Actual); Primary Completion 2016-08-24 (Actual); Study Completion 2020-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (183):
- United States (4):
  - Cancer Center of Central Connecticut, Plainville, Connecticut
  - Cancer Center of Central Connecticut, Southington, Connecticut
  - Florida Cancer Research Institute, Boca Raton, Florida
  - Florida Cancer Research Institute, Plantation, Florida
- Argentina (4):
  - COIBA - Centro de Oncologia e Investigacion Buenos Aires, Berazategui, Buenos Aires
  - Instituto De Oncologia De Rosario, Rosario, Santa Fe Province
  - Centro Medico San Roque, San Miguel de Tucumán, Tucumán Province
  - Sanatorio de la Providencia, C.a.b.a
- Brazil (11):
  - CRIO - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - Associacao de Combate ao Cancer em Goias - Hospital Araujo Jorge, Goiânia, Goiás
  - Liga Paranaense de Combate ao Cancer - Hospital Erasto Gaertner, Curitiba, Paraná
  - Instituto do Cancer de Londrina - Hospital do Cancer de Londrina - HCL, Londrina, Paraná
  - Associacao Hospital de Caridade Ijui, Ijuí, Rio Grande do Sul
  - Hospital Bruno Born (Sociedade Beneficencia e Caridade de Lajeado), Lajeado, Rio Grande do Sul
  - Centro de Pesquisa em Oncologia - Uniao Brasileira de Educacao e Assistencia, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisas Oncologicas de Santa Catarina - CEPON, Florianópolis, Santa Catarina
  - Centro de Novos Tratamentos Itajai - Clinica de Neoplasias Litoral, Itajaí, Santa Catarina
  - Fundacao Pio XII - Hospital de Cancer de Barretos, Barretos, São Paulo
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia - Faculdade de Medicina do ABC, Santo André, São Paulo
- Chile (8):
  - Clinica Alemana de Temuco, Temuco, Región de la Araucanía
  - Centro de Investigacion Clinica SIM, Temuco, Región de la Araucanía
  - Administrative office, Temuco, Región de la Araucanía
  - Hospital Clinico Vina Del Mar, Viña del Mar, Región de Valparaíso
  - Instituto Oncologico, Clinica Renaca, Viña del Mar, Región de Valparaíso
  - Fresenius Kabi Chile Therapia iv, Santiago, RM
  - Hospital Naval Almirante Nef, V Region
  - Instituto Oncologico Clinica Renaca, V Region
- Onkologicka klinika VFN a 1. LF UK, Fakultni poliklinika, Prague, Czechia
- Greece (3):
  - General Hospital of Chania "O Agios Georgios", Chania, Crete
  - Interbalkan European Medical Center, Pylaia, Thessaloniki
  - General Hospital of Athens "Hippokration", Athens
- Hungary (4):
  - Bacs-Kiskun Megyei Korhaz, Onkoradiologiai Kozpont, Kecskemét
  - Borsod-Abauj-Zemplen Megyei Korhaz, es Egyetemi Oktatokorhaz, Klinikai Onkologiai es Sugarterapias, Miskolc
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz - Rendelointezet, Megyei Onkologiai Kozpont, Szolnok
  - Markusovszky Egyetemi Oktatokorhaz, Szombathely
- India (13):
  - Department of Medicine New Block, Visakhapatnam, Andhra Pradesh
  - Manipal Hospital, Bengaluru, Karnataka
  - Manipal Centre for Clinical Research, Manipal, Karnataka
  - Tata Memorial Centre, Tata Memorial Hospital, Mumbai, Maharashtra
  - Shatabdi Super Speciality Hospital, Nashik, Maharashtra
  - Advanced Centre for Treatment Research and Education in Cancer (ACTREC), Navi Mumbai, Maharashtra
  - Deenanath Mangeshkar Hospital & Research Centre, Pune, Maharashtra
  - Sahyadri Clinical Research & Development Centre, Pune, Maharashtra
  - Sahyadri Speciality Hospital, Pune, Maharashtra
  - Acharya Harihar Regional Cancer Center, Cuttack, Odisha
  - Acharya Tulsi Regional Cancer Treatment and Research Institute, Bikaner, Rajasthan
  - Meenakshi Mission Hospital and Research Centre, Madurai, Tamil Nadu
  - MNJ Institute of Oncology & Regional Cancer Center, Hyderabad, Telangana
- Japan (15):
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Japan Community Health care Organization Kurume General Hospital, Kurume, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Saitama Cancer Center Hospital, Kitaadachi-gun, Saitama
  - Tokyo Metropolitan Cancer and Infectious diseases Center Komagome Hospital, Bunkyo-ku, Tokyo
  - National Hospital Organization Tokyo Medical Center, Meguro-Ku, Tokyo
  - Showa University Hospital, Shinagawa-ku, Tokyo
  - Chiba Cancer Center, Chiba
  - Hakuaikai Medical Corporation Sagara Hospital, Kagoshima
  - Niigata Cancer Center Hospital, Niigata
  - Nakanoshima Osaka Breast Clinic, Osaka
  - Osaka Breast Clinic, Osaka
  - Shizuoka General Hospital, Shizuoka
- P.Stradins Clinical University Hospital, Riga, Latvia
- Mexico (5):
  - Consultorio dentro de la Torre Medica Dalinde (Oncologia Medica), Mexico City, Mexico City
  - Inter Hosp S.A. de C.V. "Centro Medico Dalinde", Mexico City, Mexico City
  - Instituto Nacional de Cancerologia, Mexico City, Mexico City
  - Oaxaca Site Management Organization S.C., Oaxaca City
  - Cancerologia de Queretaro S.C., Querétaro
- Peru (8):
  - Hospital Militar Central, Lima
  - INNPARES, Lima
  - Resocentro, Lima
  - Clinica Anglo Americana, Lima
  - Instituto de Oncologia y Radioterapia de la Clinica Ricardo Palma, Lima
  - Radiologos S.R.L., Lima
  - Instituto Nacional de Enfermedades Neoplasicas, Lima
  - Siglo XXI, Lima
- Philippines (9):
  - Cebu Doctors' University Hospital, Cebu City, CEBU
  - The Research Institute at Perpetual Succor Hospital, Cebu City, Central Visayas
  - Cardinal Santos Medical Center, San Juan City, Mentro Manila
  - Manila Doctors Hospital, Manila, National Capital Region
  - Veterans Memorial Medical Center, Quezon City, National Capital Region
  - University of Philippines Manila-Philippine General Hospital, Manila, NCR
  - The Medical City, Pasig, NCR
  - St. Luke's Medical Center, Quezon City, NCR
  - Manila Doctors Hospital, Manila
- Poland (6):
  - COPERNICUS Podmiot Leczniczy Sp. z o.o. Wojewodzkie Centrum Onkologii, Gdansk
  - Szpitale Pomorskie Sp. z o.o. Oddzial Onkologii i Radioterapii, Gdynia
  - Centrum Terapii Wspolczesnej, Lodz
  - SPZOZ MSW z Warminsko-Mazurskim Centrum Onkologii w Olsztynie, Oddzial Kliniczny Chemioterapii, Olsztyn
  - MRUKMED. Lekarz Beata Madej Mruk i Partner. Sp. p. Oddzial nr 1 w Rzeszowie, Rzeszów
  - Magodent Sp. z o.o. Oddzial Onkologii Klinicznej/Chemioterapii, Warsaw
- Portugal (2):
  - Hospital de Braga, Braga
  - Hospital CUF Descobertas, Lisbon
- Romania (8):
  - Institutul Oncologic Prof. Dr. Ion Chiricuta, Cluj-Napoca, Cluj
  - S.C. Medisprof S.R.L, Cluj-Napoca, Cluj
  - Centrul de Oncologie Sf. Nectarie, Craiova, Dolj
  - SC Oncolab SRL, Oncologie, Craiova, JUD DOLJ
  - Spitalul Universitar de Urgenta, Departamentul Oncologie Medicala, Bucharest
  - Spitalul Clinic Judetean de Urgenta Sibiu, Sibiu
  - Spitalul Judetean de Urgenta "Sf.Ioan cel Nou", Sectia Oncologie, Suceava
  - Spitalul Clinic Municipal de Urgenta Timisoara, Sectia Clinica Oncologie Medicala, Timișoara
- Russia (39):
  - GBUZ Republican Clinical Hospital n.a. G.F. Kuvatova, Ufa, Bashkortostan Republic
  - Republican Clinical Oncology Dispensary of the Ministry of Healthcare of Baskortostan Republic, Ufa, Bashkortostan Republic
  - State Healthcare Institution, Republican Clinical Oncology Dispensary of the Ministry of, Ufa, Bashkortostan Republic
  - Republic Clinical Hospital of Emergency Care, Grozny, Chechenkaya Republic
  - State Healthcare Institution Kursk Regional Oncological Dispensary of the Healthcare Committee, Kislino Settlement, Kursk Oblast
  - State Budgetary Healthcare Institution "Leningrad Regional Oncological Dispensary", Kuzmolovo, Vsevolozhskiy, Leningradskaya Oblast'
  - FSBSI Russian Cancer Research Center n.a. N.N.Blokhin, Moscow, NAP
  - GBUZ of Perm region "Perm regional oncology dispensary", Perm, NAP
  - Federal State Budgetary Institution ¿National Medical Research Oncology Centre named after N.N., Saint Petersburg, Pos.pesochny
  - State Budgetary Healthcare Institution ''Republic Oncological Dispensary'', Petrozavodsk, Republic of Karelia
  - State budget institution of healthcare of Mordovia Republic "Republic Oncology Dispensary", Saransk, Respublika Mordoviya
  - Rostov Research Institute of Oncology, Rostov-on-Don, Rostov Oblast
  - Saint-Petersburg Clinical Research Center of Specialized Types of Medical Care (Oncology), Poselok Pesochny, Sankt-Peterburg
  - Private medical institution Euromedservice, Pushkin, Sankt-Peterburg
  - LLC Medekspert, Kislovodsk, Stavropol Kray
  - Federal State Budgetary Healthcare Institution of "Clinical Hospital #101 of Federal Medical and, Lermontov, Stavropol Kray
  - Centre of Specialized kinds of Medical Care of Pyatigorsk city, Pyatigorsk, Stavropol Kray
  - State Budgetary Healthcare Institution of Stavropol Region Pyatigorsk Oncology Dispensary, Pyatigorsk, Stavropol Kray
  - LLC Novaya Clinica, Pyatigorsk, Stavropol Kray
  - Pyatigorsk City Hospital #2, Pyatigorsk, Stavropol Kray
  - Stavropol Regional Hospital for War Veterans, Pyatigorsk, Stavropol Kray
  - State Budgetary Healthcare Institution Volgograd Regional Clinical Oncology Dispensary, Volzhsky, Volgograd Oblast
  - GBUZ Arkhangelsk Regional Clinical Oncological dispensary, Arkhangelsk
  - State Budgetary Healthcare Institution "Chelyabinsk Regional Clinical Oncological Dispensary", Chelyabinsk
  - "Regional Budgetary Healthcare Institution ""Ivanovo Regional Oncology Dispensary""", Ivanovo
  - SBIH of Kaluga Region "Kaluga Regional Clinical Oncology Dispensary", Kaluga
  - GBUZ "Regional Oncology Dispensary #2", Magnitogorsk
  - Federal State Budgetary Institution "Russian Oncological Scientific Center n.a. N.N. Blokhin" of, Moscow
  - LLC VitaMed, Moscow
  - State Budgetary Healthcare Institution "Nizhniy Novgorod Regional Oncological Dispensary", Nizhny Novgorod
  - "BIH of Omsk Region ""Clinical oncological dispensary""", Omsk
  - Budgetary Institution of Healthcare of Orel region "Orel oncological dispensary", Oryol
  - SBEI HPE RyazSMU of MoH of the Russian Federation based on SBI of Ryazan Region "Regional CLinical, Ryazan
  - SBI "North-Western State Medical University n.a. I. I. Mechnikov" of the MoH of the Russian, Saint Petersburg
  - Non-state healthcare agency Road Clinical Hospital PLC Russian Railways, Saint Petersburg
  - Saint-Petersburg State Budgetary Healthcare Institution "Oncological Dispensary of Moscow District", Saint Petersburg
  - SBEI of HPE "First Saint Petersburg State Medical University, Saint Petersburg
  - Non-State Healthcare Institution "Road Clinical Hospital at Saratov II Station", Saratov
  - State Budgetary Healthcare Institution of Stavropol region "Stavropol regional clinical oncology, Stavropol
- Serbia (4):
  - Institute for Oncology and Radiology of Serbia, Belgrade
  - Military Medical Academy, Belgrade
  - Oncology Institute of Vojvodina, Kamenitz
  - Clinic of Oncology-Clinical Center Nis, Niš
- Slovakia (2):
  - Onkologicky ustav sv. Alzbety, s.r.o., Bratislava
  - Narodny Onkologicky Ustav, Bratislava
- South Africa (8):
  - GVI Oncology, Langenhoven Drive Oncology Centre, Port Elizabeth, Eastern Cape
  - wits Clinical Research, Joannesburg, Gauteng
  - The Medical Oncology Centre of Rosebank, Johannesburg, Gauteng
  - Sandton Oncology Centre, Johannesburg, Gauteng
  - *Department of Medical Oncology, University of Pretoria & Steve Biko Academic Hospitals Complex, Pretoria, Gauteng
  - Eastleigh Breast Care Centre, Pretoria, Gauteng
  - Cape Town Oncology Trials, Kraaifontein, Western Cape
  - GVI Rondebosch Oncology Centre-Rondebosch Medical Centre, Rondebosch, Western Cape
- South Korea (8):
  - Ulsan University Hospital, Ulsan, Korea
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Pusan National University Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - National Cancer Centre, Goyang-si
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Korea University Guro Hospital, Seoul
- Thailand (3):
  - National Cancer Institute, Ratchathewi, Bangkok
  - Udonthani Cancer Hospital, Amphur Muang, Udonthani
  - Faculty of Medicine, Chulongkorn University, Medical Oncology Unit, Bangkok
- Turkey (Türkiye) (6):
  - Baskent University School of Medicine Adana Hospital, Adana
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Uludag Universitesi Tip Fakultesi Ic Hastaliklari Anabilim Dali, Bursa
  - Dicle University Medical Faculty, Diyarbakır
  - Gaziantep University Medical Faculty, Gaziantep
  - Istanbul Universitesi Onkoloji Enstitusu, Istanbul
- Ukraine (11):
  - Municipal Institution "Chernivtsi Regional Clinical Oncology Center", Outpatient Department, Chernivtsi
  - Municipal Non-Profit Enterprise City Clinical Hospital No.4of Dnipro Regional Council, Department of, Dnipro
  - SI Institute of Medical Radiology n.a.S.P. Ilrygoriev of National Academy of Medical Science of, Kharkiv
  - Communal Non-Profit Enterprise "Regional Center of Oncology", Kharkiv
  - Khmelnytskyi Regional Oncologic Dispensary, Khmelnytskyi
  - Municipal Enterprise 'Kryvyi Rih Oncology Dispensary of Dnipropetrovsk Regional Council', Kryvyi Rih
  - Municipal Non-Profit Enterprise of Kyiv Regional Council "Kyiv Regional Oncology Dispensary", Kyiv
  - Lviv State Oncologic Regional Treatment and Diagnostic Center, Lviv
  - Municipal Institution Odesa Regional Clinical Hospital, Mammology Center, Odesa
  - Zakarpattia Regional Clinical Oncological Center, Uzhhorod
  - Municipal Non-profit Enterprise Podilsk Regional Oncology Centre of Vinnytsia Regional Council, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Li RK, Tokunaga E, Adamchuk H, Vladimirov V, Yanez E, Lee KS, Bondarenko I, Vana A, Hilton F, Ishikawa T, Tajima K, Lipatov O. Long-Term Safety and Effectiveness of PF-05280014 (a Trastuzumab Biosimilar) Treatment in Patients with HER2-Positive Metastatic Breast Cancer: Updated Results of a Randomized, Double-Blind Study. BioDrugs. 2022 Jan;36(1):55-69. doi: 10.1007/s40259-021-00513-7. Epub 2022 Feb 8. PMID 35133617
- [Derived] Chen X, Li C, Ewesuedo R, Yin D. Population pharmacokinetics of PF-05280014 (a trastuzumab biosimilar) and reference trastuzumab (Herceptin(R)) in patients with HER2-positive metastatic breast cancer. Cancer Chemother Pharmacol. 2019 Jul;84(1):83-92. doi: 10.1007/s00280-019-03850-1. Epub 2019 May 3. PMID 31053945
- [Derived] Pegram MD, Bondarenko I, Zorzetto MMC, Hingmire S, Iwase H, Krivorotko PV, Lee KS, Li RK, Pikiel J, Aggarwal R, Ewesuedo R, Freyman A, Li R, Vana A, Yin D, Zacharchuk C, Tan-Chiu E. PF-05280014 (a trastuzumab biosimilar) plus paclitaxel compared with reference trastuzumab plus paclitaxel for HER2-positive metastatic breast cancer: a randomised, double-blind study. Br J Cancer. 2019 Jan;120(2):172-182. doi: 10.1038/s41416-018-0340-2. Epub 2018 Dec 20. PMID 30568294
- See also: Related Info — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3271002&StudyName=A%20Phase%203%20Randomized%2C%20Double-blind%20Study%20Of%20Pf-05280014%20Plus%20Paclitaxel%20Versus%20Trastuzumab%20Plus%20Paclitaxel%20For%20The%20First-line%20Treatment%20Of%20Patients%20With%20Her2-positive%20Metastatic%20Breast%20Cancer

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 707 participants were randomized to the study. Of these, 5 participants were randomized but did not receive the study drug.
Pre-assignment Details: Participants who fulfilled the inclusion/exclusion criteria were randomly assigned to 1 of the 2 treatments of this study.
Groups:
- PF-05280014: Participants with human epidermal growth factor receptor 2 (HER2)-positive breast cancer received PF-05280014 on Days 1, 8, 15 and 22 of each 28-day cycle followed by paclitaxel on Days 1, 8 and 15 of each 28-day cycle both as intravenous (IV) infusions until the end of the study. The first infusion of PF-05280014 was 4 mg/kg over 90 minutes on Cycle 1 Day 1. Subsequent weekly infusions of PF-05280014 were 2 mg/kg over 30 to 90 minutes. Paclitaxel was administered at a dose of 80 mg/m^2 over 60 minutes. Following completion of the paclitaxel administration period and beginning no earlier than Week 33 of the study, the PF-05280014 could be changed at the discretion of the investigator to every 3 weeks at a dose of 6 mg/kg infused over 30 to 90 minutes depending on tolerability.
- Trastuzumab-EU: Participants with HER2-positive breast cancer received trastuzumab-EU on Days 1, 8, 15 and 22 of each 28-day cycle followed by paclitaxel on Days 1, 8 and 15 of each 28-day cycle both as IV infusions until the end of the study. The first infusion of trastuzumab-EU was 4 mg/kg over 90 minutes on Cycle 1 Day 1. Subsequent weekly infusions of trastuzumab-EU were 2 mg/kg over 30 to 90 minutes. Paclitaxel was administered at a dose of 80 mg/m^2 over 60 minutes. Following completion of the paclitaxel administration period and beginning no earlier than Week 33 of the study, the trastuzuamab-EU could be changed at the discretion of the investigator to every 3 weeks at a dose of 6 mg/kg infused over 30 to 90 minutes depending on tolerability.
Period: Overall Study
Arm/Group | PF-05280014 | Trastuzumab-EU
Started | 352 | 355
Treated | 349 | 353
Completed | 234 | 217
Not Completed | 118 | 138
Not completed — Death | 52 | 60
Not completed — Protocol Violation | 2 | 1
Not completed — Lost to Follow-up | 8 | 18
Not completed — No longer willing to participate in study | 26 | 26
Not completed — Participants terminated from study by Sponsor | 26 | 30
Not completed — Other | 4 | 3

BASELINE CHARACTERISTICS:
Population: The baseline analysis population was based on the safety population, which was defined as all participants who were randomized and treated with study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-05280014 | Trastuzumab-EU | Total
Number analyzed (Participants) | 349 | 353 | 702
Age, Customized [Number; unit: Participants]
  <18 | 0 | 0 | 0
  18 to 64 | 283 | 292 | 575
  65 to 84 | 66 | 60 | 126
  ≥85 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 349 | 353 | 702
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Derived From Central Radiology Assessments: ITT Population
Description: ORR was defined as the percentage of participants who achieved complete response (CR, complete disappearance of all target lesions with the exception of nodal disease; all target nodes must have decreased to normal size [short axis <10 mm]) or partial response (PR, >=30% decrease from baseline of the sum of diameters (SOD) of all target measurable lesions; the short diameter was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions) by Week 25 of the study and confirmed on a follow-up assessment (Week 33+/-14 days), based on the assessments of the central radiology review in accordance with RECIST 1.1.
Time Frame: From the date of randomization until all participants had either completed the Week 33 tumor assessment or discontinued study drug earlier than the Week 33 visit
Population: The ITT population was defined as all participants who were randomized to study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-05280014 | Trastuzumab-EU
Number analyzed (Participants) | 352 | 355
percentage of participants | 62.5 [57.2 to 67.6] | 66.5 [61.3 to 71.4]
Statistical Analysis 1: Comparison: PF-05280014 vs Trastuzumab-EU; Risk Ratio and associated 95% confidence interval (CI) are unstratified and based on the Miettinen and Nurminen method; Test type: Equivalence — The hypothesis to be tested in this study was that the risk ratio of ORR of PF-05280014 versus that of trastuzumab-EU by Week 25 (+/-14 days) was within a pre-specified margin of 0.80 to 1.25; Risk Ratio (RR) = 0.940, 95% CI 2-sided [0.842 to 1.049]

2. Secondary Outcome: One-year Progression-Free Survival (PFS) Rate Derived From Central Radiology Assessments: ITT Population
Description: One-year PFS rate was analyzed based on the time from date of randomization to first documentation of progressive disease (PD), or death due to any cause in the absence of documented PD, based on the assessments of the central radiology review in accordance with RECIST 1.1. PD was defined for target disease as at least a 20% increase in sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum was observed during therapy) with a minimum absolute increase of 5 mm. For non-target disease: PD was defined as unequivocal progression of pre-existing lesions and if overall tumor burden increased sufficiently to merit discontinuation of therapy; appearance of any new unequivocal malignant lesion was also considered PD. The 95% CI for the median time to event was based on the Brookmeyer and Crowley method.
Time Frame: From the date of randomization until 378 days post-randomization
Population: The ITT population was defined as all participants who were randomized to study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PF-05280014 | Trastuzumab-EU
Number analyzed (Participants) | 352 | 355
months | 12.16 [11.93 to 12.48] | 12.06 [11.79 to NA] — There are insufficient events to estimate the upper bound of the 95% CI.
Statistical Analysis 1: Comparison: PF-05280014 vs Trastuzumab-EU; Test type: Superiority; p = 0.505, Log Rank — 1-sided log-rank test was used to compare the PFS distribution between the two treatment groups and was stratified by prior trastuzumab exposure (Yes/No) and estrogen receptor (ER) status (ER positive vs. ER negative); Cox Proportional Hazard = 1.00, 95% CI 2-sided [0.80 to 1.26] — The 95% CI for the hazard ratio was based on the Cox's proportional hazard model

3. Secondary Outcome: Duration of Response (DOR) Per Central Radiology Assessments: ITT Population
Description: DOR:time from first documentation of objective response (CR or PR) to first documentation of PD/death due to any cause in absence of documented PD, based on central radiology review. As per RECIST v1.1, CR:complete disappearance of all target lesions with exception of nodal disease; all target nodes reduced in short axis <10 mm. PR: >=30% decrease from baseline of SOD of target lesions; short diameter used in sum for target nodes,longest diameter used in sum for other target lesions. PD for target disease:at least 20% increase in SOD of target lesions above smallest sum observed (over baseline if no decrease in sum observed) with minimum absolute increase of 5 mm. For non-target disease:unequivocal progression of pre-existing lesions and if overall tumor burden increased sufficiently to merit discontinuation of therapy; appearance of any new unequivocal malignant lesion was also considered PD. The 95% CI for median time to event was based on the Brookmeyer and Crowley method.
Time Frame: From the date of randomization until 378 days post-randomization
Population: The ITT population was defined as all participants who were randomized to study drug. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PF-05280014 | Trastuzumab-EU
Number analyzed (Participants) | 224 | 238
months | 11.27 [10.41 to 11.27] | 10.58 [10.22 to NA] — There are insufficient events to estimate the upper bound of the 95% CI.
Statistical Analysis 1: Comparison: PF-05280014 vs Trastuzumab-EU; Test type: Superiority; p = 0.304, Log Rank — 1-sided log-rank test was used to compare the DOR distribution between the two treatment groups and was stratified by prior trastuzumab exposure (Yes/No) and ER status (ER positive vs. ER negative); Cox Proportional Hazard = 0.92, 95% CI 2-sided [0.67 to 1.27] — The 95% CI for the hazard ratio was based on the Cox's proportional hazard model

4. Secondary Outcome: Overall Survival: ITT Population
Description: Overall survival was analyzed based on the time from date of randomization to the date of death due to any cause. Participants last known to be alive were censored on the date of last contact. The 95% CI for the median time to event was based on the Brookmeyer and Crowley Method.
Time Frame: From the date of randomization until end of study (approximately 6 years)
Population: The ITT population was defined as all participants who were randomized to study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PF-05280014 | Trastuzumab-EU
Number analyzed (Participants) | 352 | 355
months | NA [NA to NA] — There were insufficient events to estimate the median survival and the 95% CI. | NA [NA to NA] — There were insufficient events to estimate the median survival and the 95% CI.
Statistical Analysis 1: Comparison: PF-05280014 vs Trastuzumab-EU; Test type: Superiority; p = 0.339, Log Rank — 1-sided log-rank test was used to compare the OS distribution between the two treatment groups and was stratified by prior trastuzumab exposure (Yes/No) and ER status (ER positive vs. ER negative); Cox Proportional Hazard = 0.929, 95% CI 2-sided [0.656 to 1.316] — The 95% CI for the hazard ratio was based on the Cox's proportional hazard model

5. Secondary Outcome: Serum Peak Concentration of PF-05280014 at Selected Cycles: Pharmacokinetics (PK) Population
Description: Human PK serum samples were analyzed for concentrations of PF-05280014 using a validated, sensitive, and specific enzyme-linked immunosorbent assay (ELISA).
Time Frame: 1 hour post end of infusion on Day 1 of Cycles 1 and 5
Population: PK population was used for analysis, included all participants who received PF-05280014 or trastuzumab-EU and had no major protocol deviations that influenced PK assessments, and had at least 1 post dose concentration measurement. Here "number analyzed (n)" signifies participants evaluable at specified time points only.
Measure: Median (Full Range); unit: mcg/mL
Arm/Group | PF-05280014
Number analyzed (Participants) | 349
mcg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 278
  Cycle 1 Day 1 | 89.85 [0.00 to 246]
  Cycle 5 Day 1: number analyzed (Participants) | 204
  Cycle 5 Day 1 | 95.70 [0.00 to 435]

6. Secondary Outcome: Serum Peak Concentration of Trastuzumab-EU at Selected Cycles: PK Population
Description: Human PK serum samples were analyzed for concentrations of trastuzumab-EU using a validated, sensitive, and specific ELISA.
Time Frame: 1 hour post end of infusion on Day 1 of Cycles 1 and 5
Population: PK population was used for analysis, included all participants who received PF-05280014 or trastuzumab-EU and had no major protocol deviations that influenced PK assessments, and had at least 1 post dose concentration measurement. Here "n" signifies participants evaluable at specified time points only.
Measure: Median (Full Range); unit: mcg/mL
Arm/Group | Trastuzumab-EU
Number analyzed (Participants) | 353
mcg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 267
  Cycle 1 Day 1 | 89.70 [0.00 to 273]
  Cycle 5 Day 1: number analyzed (Participants) | 221
  Cycle 5 Day 1 | 94.40 [8.96 to 353]

7. Secondary Outcome: Serum Trough (Pre-dose) Concentration of PF-05280014 at Selected Cycles: PK Population
Description: Human PK serum samples were analyzed for concentrations of PF-05280014 using a validated, sensitive, and specific ELISA.
Time Frame: Pre-dose on Day 1 of Cycles 1, 3, 4, 5, 7, 8, 11, 14, 17 and Day 8 of Cycles 1 and 5
Population: PK population.Here "n" signifies participants evaluable at specified time points only.The Cycle 17 Day 1 (C17D1) samples summarized previously at PCD (Week 33) fell outside of cut-off used for final analysis (Week 53), to limit data for up to 1-year post randomization, which was more conservative from previous Week 33 analysis. While comparing data between Week 33 and Week 53, there was a significant drop off in number of samples summarized at C17D1 and was down to zero for this outcome measure.
Measure: Median (Full Range); unit: mcg/mL
Arm/Group | PF-05280014
Number analyzed (Participants) | 349
mcg/mL
  Cycle 1 Day 1 | 0.00 [0.00 to 123]
  Cycle 1 Day 8: number analyzed (Participants) | 339
  Cycle 1 Day 8 | 27.90 [0.00 to 91.5]
  Cycle 3 Day 1: number analyzed (Participants) | 309
  Cycle 3 Day 1 | 48.20 [0.00 to 110]
  Cycle 4 Day 1: number analyzed (Participants) | 304
  Cycle 4 Day 1 | 53.50 [0.00 to 150]
  Cycle 5 Day 1: number analyzed (Participants) | 288
  Cycle 5 Day 1 | 57.00 [0.00 to 182]
  Cycle 5 Day 8: number analyzed (Participants) | 277
  Cycle 5 Day 8 | 57.40 [9.85 to 174]
  Cycle 7 Day 1: number analyzed (Participants) | 265
  Cycle 7 Day 1 | 60.50 [0.00 to 152]
  Cycle 8 Day 1: number analyzed (Participants) | 256
  Cycle 8 Day 1 | 62.25 [0.00 to 140]
  Cycle 11 Day 1: number analyzed (Participants) | 220
  Cycle 11 Day 1 | 54.65 [0.00 to 148]
  Cycle 14 Day 1: number analyzed (Participants) | 188
  Cycle 14 Day 1 | 50.70 [0.00 to 189]
  Cycle 17 Day 1: number analyzed (Participants) | 0

8. Secondary Outcome: Serum Trough (Pre-dose) Concentration of Trastuzumab-EU at Selected Cycles: PK Population
Description: as for outcome 6
Time Frame: Pre-dose on Day 1 of Cycles 1, 3, 4, 5, 7, 8, 11, 14, 17 and Day 8 of Cycles 1 and 5
Population: as for outcome 6
Measure: Median (Full Range); unit: mcg/mL
Arm/Group | Trastuzumab-EU
Number analyzed (Participants) | 353
mcg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 349
  Cycle 1 Day 1 | 0.00 [0.00 to 98.0]
  Cycle 1 Day 8: number analyzed (Participants) | 340
  Cycle 1 Day 8 | 29.80 [0.00 to 101]
  Cycle 3 Day 1: number analyzed (Participants) | 319
  Cycle 3 Day 1 | 50.40 [1.74 to 171]
  Cycle 4 Day 1: number analyzed (Participants) | 316
  Cycle 4 Day 1 | 54.35 [0.00 to 148]
  Cycle 5 Day 1: number analyzed (Participants) | 303
  Cycle 5 Day 1 | 60.00 [0.00 to 244]
  Cycle 5 Day 8: number analyzed (Participants) | 287
  Cycle 5 Day 8 | 61.20 [4.64 to 150]
  Cycle 7 Day 1: number analyzed (Participants) | 276
  Cycle 7 Day 1 | 63.00 [1.93 to 340]
  Cycle 8 Day 1: number analyzed (Participants) | 262
  Cycle 8 Day 1 | 65.55 [0.690 to 155]
  Cycle 11 Day 1: number analyzed (Participants) | 223
  Cycle 11 Day 1 | 57.50 [1.52 to 251]
  Cycle 14 Day 1: number analyzed (Participants) | 173
  Cycle 14 Day 1 | 54.60 [0.00 to 187]
  Cycle 17 Day 1: number analyzed (Participants) | 1
  Cycle 17 Day 1 | 45.10 [45.1 to 45.1]

9. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADA) Sample: Safety Population
Description: Two sensitive, specific, and semi-quantitative electrochemiluminescent (ECL) immunoassays, 1 for detecting antibodies against PF-05280014 and the other for detecting antibodies against trastuzumab, were used to analyze ADA samples. Serum samples were first screened for ADA. Any samples that were positive in the screening assay were further analyzed to confirm the positive result and determine the antibody titers. All samples were taken prior to dosing. The number of participants with a positive sample (titer >=1.0) is provided.
Time Frame: Pre-dose on Day 1 of Cycles 1, 3, 5, 8, 11, 14, 17
Population: Safety population was used for analysis, included all participants who received at least 1 dose of study drug. Here "n" signifies participants evaluable at specified time points only.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-05280014 | Trastuzumab-EU
Number analyzed (Participants) | 349 | 353
Participants
  Cycle 1 Day 1 (prior to treatment): number analyzed (Participants) | 349 | 350
  Cycle 1 Day 1 (prior to treatment) | 30 | 14
  Cycle 3 Day 1: number analyzed (Participants) | 308 | 321
  Cycle 3 Day 1 | 0 | 0
  Cycle 5 Day 1: number analyzed (Participants) | 287 | 303
  Cycle 5 Day 1 | 0 | 0
  Cycle 8 Day 1: number analyzed (Participants) | 255 | 263
  Cycle 8 Day 1 | 0 | 0
  Cycle 11 Day 1: number analyzed (Participants) | 223 | 224
  Cycle 11 Day 1 | 0 | 0
  Cycle 14 Day 1: number analyzed (Participants) | 192 | 175
  Cycle 14 Day 1 | 0 | 0
  Cycle 17 Day 1: number analyzed (Participants) | 0 | 1
  Cycle 17 Day 1 |  | 0

10. Secondary Outcome: Number of Participants With Positive Neutralizing Antibodies (Nab) Prior to Treatment: Safety Population
Description: Human serum samples testing positive for the presence of ADA (anti-PF-05280014 or anti-trastuzumab-EU) were analyzed for the presence or absence of NAb (neutralizing anti-PF-05280014 or neutralizing anti-trastuzumab-EU antibodies) following a tiered approach using screening and titer determination. The number of participants at baseline (prior to treatment) with a positive NAb sample (titer >=1.48) is provided.
Time Frame: Cycle 1 Day 1 (prior to treatment)
Population: Safety population was used for analysis, included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-05280014 | Trastuzumab-EU
Number analyzed (Participants) | 349 | 350
Participants | 20 | 9

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious AEs (SAEs) which occurred from the time the participant had taken at least 1 dose of study drug and the time of informed consent, respectively, through 70 days after the last dose of study drug (maximum up to 328 weeks)
Description: All-cause mortality: The total number of deaths occurred during study are reported for all randomized participants, not only for treated participants, and included deaths which occurred beyond 70 days post last study drug dose (i.e. beyond 328 weeks). SAEs and other AEs: Analysis performed on safety population. The safety population included all participants who received at least 1 dose of study drug.
Arm/Group | PF-05280014 | Trastuzumab-EU
All-Cause Mortality (participants affected / at risk) | 61/349 | 67/353
Serious Adverse Events (participants affected / at risk) | 67/349 | 69/353
Other Adverse Events (participants affected / at risk) | 337/349 | 334/353
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-05280014 (N=349) | Trastuzumab-EU (N=353)
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 4
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Macular degeneration (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Proctalgia (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Cyst rupture (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Disease progression (General disorders) | 15 | 16
Fatigue (General disorders) | 1 | 1
Pyrexia (General disorders) | 0 | 4
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 4
Cystitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Mastitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 6 | 3
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 2
Septic shock (Infections and infestations) | 2 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 2
Wound infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1
Ejection fraction decreased (Investigations) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 3
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 3 | 0
Vocal cord paralysis (Nervous system disorders) | 1 | 0
Affective disorder (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 2
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0
Embolism (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Thyroiditis subacute (Endocrine disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Infected skin ulcer (Infections and infestations) | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nasopharyngeal neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Cerebral venous sinus thrombosis (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-05280014 (N=349) | Trastuzumab-EU (N=353)
Anaemia (Blood and lymphatic system disorders) | 122 | 134
Leukopenia (Blood and lymphatic system disorders) | 36 | 45
Neutropenia (Blood and lymphatic system disorders) | 97 | 94
Abdominal pain (Gastrointestinal disorders) | 14 | 32
Constipation (Gastrointestinal disorders) | 24 | 31
Diarrhoea (Gastrointestinal disorders) | 61 | 65
Nausea (Gastrointestinal disorders) | 58 | 70
Stomatitis (Gastrointestinal disorders) | 23 | 13
Vomiting (Gastrointestinal disorders) | 28 | 26
Asthenia (General disorders) | 53 | 46
Fatigue (General disorders) | 46 | 51
Oedema peripheral (General disorders) | 27 | 45
Pyrexia (General disorders) | 41 | 29
Respiratory tract infection viral (Infections and infestations) | 23 | 13
Upper respiratory tract infection (Infections and infestations) | 36 | 46
Infusion related reaction (Injury, poisoning and procedural complications) | 33 | 31
Alanine aminotransferase increased (Investigations) | 42 | 45
Aspartate aminotransferase increased (Investigations) | 36 | 31
Blood alkaline phosphatase increased (Investigations) | 28 | 26
Ejection fraction decreased (Investigations) | 49 | 45
Weight increased (Investigations) | 20 | 22
Decreased appetite (Metabolism and nutrition disorders) | 23 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 44 | 38
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 33
Bone pain (Musculoskeletal and connective tissue disorders) | 20 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 26 | 35
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 | 24
Dizziness (Nervous system disorders) | 38 | 30
Headache (Nervous system disorders) | 53 | 73
Neuropathy peripheral (Nervous system disorders) | 33 | 34
Peripheral sensory neuropathy (Nervous system disorders) | 93 | 85
Cough (Respiratory, thoracic and mediastinal disorders) | 33 | 32
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 22
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15 | 23
Alopecia (Skin and subcutaneous tissue disorders) | 189 | 186
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 23
Rash (Skin and subcutaneous tissue disorders) | 26 | 26
Hypertension (Vascular disorders) | 40 | 33
Thrombocytopenia (Blood and lymphatic system disorders) | 18 | 12
Dyspepsia (Gastrointestinal disorders) | 16 | 18
Chills (General disorders) | 17 | 18
Nasopharyngitis (Infections and infestations) | 21 | 19
Urinary tract infection (Infections and infestations) | 5 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.